CLINICAL TRIAL: NCT00690664
Title: Evaluation of Scalp and Hair Shaft With Biologic Markers in African American and Caucasian Hair
Status: Completed | Type: Observational
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: IRB00002509; 31716
Record Dates: First submitted 2008-06-02; First posted 2008-06-05 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Scalp Health
Keywords: Hair characteristics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Hair, both broken strands and those that release from the scalp with bulb intact.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- B: Caucasian women
- A: African American women

SUMMARY:
The purpose of this research study is to better understand African American hair and scalp, its biologic appearance and how this relates to African Americans' perceptions of their hair and scalp health. Since most hair studies have looked at Caucasian hair and scalp, we will use a population of Caucasian subjects for comparison in evaluating various hair and scalp parameters.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing to sign informed consent
* Female from the ages of 21-60 years
* Must be willing to have a thorough scalp and hair shaft examination
* Must be willing to discuss hair care regimen currently and in the past
* Must have washed hair at least 48 hours prior to initial study visit
* Pregnant and nursing females will not be allowed in the study; a baseline pregnancy test will be done to exclude pregnancy on females of childbearing potential
* Must be >6 months (26 weeks) postpartum
* Must have sufficient contrast between scalp skin color and hair color
* Must have hair at least 2 inches long
* May have mild itching and mild scaling of the scalp
* Must be willing to have hair clipped and shaved to 1mm within an approximately 2.5cm test site
* Must be in good stable general health, with no current infections.

Exclusion Criteria:

* May not have sewn-in or glued hair pieces or extensions at the time of the study
* Must not cut hair during the study
* Must not have hair loss beyond what is considered normal in the opinion of the Investigator at the time of the study
* Must not color hair or have other salon-type procedures (relaxer, permanent, highlighting, etc.) performed within 2 weeks of the initial visit
* Must not have any other underlying scalp disorder that could interfere with the test procedures or findings
* Must not have lost ≥10% of body weight within the past 12 months
* Must not have been on a weight reduction program overseen by a physician or nutritionist within the past 12 months
* Has used hair growth products e.g. minoxidil in the past 18 months
* Has undergone a hair transplant or scalp reduction surgery
* Has participated in a hair growth study within the past 15 months
* Is currently participating in another clinical study at this or any other facility
* Is taking, for a chronic condition, any prescription or over the counter medication(s) that in the opinion of the Investigator are likely to affect the hair properties (e.g. immunosuppressive agents, corticosteroids; or chronic use of anti-inflammatory medication)
* Application of any over-the-counter or prescription drug to the scalp on a routine basis within the past 3 months including but not limited to retinoids (e.g. retinal, tretinoin, retinyl palmitate, retinyl acetate, retinyl propionate), topical corticosteroids, benzyl peroxide, or any topical hormone therapy (e.g. Eterna 27)

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy female subjects between the ages of 21-60 will be enrolled in this study. These subjects will be recruited from Wake Forest University Health Sciences Dermatology clinic and our Institutional Review Board (IRB) approved advertising. Half of the participants will be African American and the other half will be Caucasian.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-04-24 (Actual); Primary Completion 2014-07-14 (Actual); Study Completion 2014-07-14 (Actual)

PRIMARY OUTCOMES:
Observe comparators of African American and Caucasian women's hair | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Amy McMichael, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No